CLINICAL TRIAL: NCT05526092
Title: OAT-GUT-BRAIN: Comprehensive Health Effects of Long-term Consumption of Oats in Metabolically Challenged Volunteers - Gut-mediated Metabolomics and Vitality
Brief Title: OAT-GUT-BRAIN: Effects of Oats and Rice on Comprehensive Health of Metabolically Challenged Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OGB
Record Dates: First submitted 2022-08-26; First posted 2022-09-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: High Cholesterol/Hyperlipidemia; High Blood Pressure; Overweight and Obesity
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Hypertension; Overweight; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oat-rich and low-gluten diet (Experimental): Participants will consume oats and oat products and follow low-gluten diet for 6 weeks.
  Interventions: Other: Dietary intervention
- Rice-rich and low-gluten diet (Placebo Comparator): Participants will consume rice and rice products and follow low-gluten diet for 6 weeks.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Changes in metabolism, microbiota, vitality and comprehensive health after 6 week consumption of oat / rice.

SUMMARY:
The overall objective of this research entity is to reveal the holistic health impact of oats in metabolically challenged individuals in a 6-week intervention, compared to that of rice. This is achieved by investigation of the plasma lipids, plasma antioxidant status, fecal microbiota and fecal bile acids. Additionally the effect of the 6-week diet on posptprandial glycemia and postprandial satiety and vitality are investigated.

DETAILED DESCRIPTION:
Aims in this 6-week randomised, single-blinded clinical trial, including a postprandial study at the 6 week time point, with metabolically challenged volunteers on oat-rich low-gluten diet, are to:

1. Compare effect of oat and rice rich diets to blood lipid and glucose status, perceived gut well-being and diet quality.
2. Investigate changes in microbiota, SCFAs, plasma antioxidant status and inflammation markers resulting from consumption of oat or rice rich low gluten diets.
3. Examine the impact of the oat and rice rich gluten free diet on the change in metabolite profiles in blood.
4. Find out the long-term effects of oat and rice consumption on recovery and vitality by modulating the gut-brain axis and measured with neuropsychological testing and using tryptophan metabolites as markers.
5. Discover how the long-term consumption of oats and rice and their possible alterations in gut microbiota affect subsequent postprandial glycaemia and response of microbiota to the meal (as seen in plasma SCFAs).

ELIGIBILITY:
Inclusion Criteria:

* Commits to follow low-gluten diet for 6 weeks
* 30 - 68 years of age
* BMI > 25 kg/m^2
* High cholesterol AND/OR Hypertension

Exclusion Criteria:

* Regular medication that can affect the gut
* Pregnancy or lactation
* Recent course of antibiotics (less than 3 months prior to the study)

Ages: 30 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in plasma short-chain fatty acids | Week 0 and 6
  Samples are taken 90 and 180 min after consuming the study meal, and at the fasting state, before and after the 6-week diet intervention to see the change between fasting state and postprandial states.
Changes from baseline in plasma antioxidant capasity | Week 0 and 6
  Plasma samples are taken 180 min after consuming the study meal, and at the fasting state, before and after the 6-week diet intervention to see the change between fasting state and postprandial states. The antioxidant status of plasma will be analysed with commercial kits for 2,2'-azino-bis-3-ethylbenzthiazoline-6-sulfonic acid (ABTS) and Oxygen Radical Absorbance Capacity (ORAC) (Merck KGaA, Darmstadt, Germany) to measure antioxidant capacity of plasma.
Changes in blood lipid | Week 0 and 6
  Postprandial plasma samples are taken at the fasting state and 15, 30, 45, 60, 90, 120 and 180 min after consuming the study meal before, and after the 6-week diet intervention to see blood lipid development curve in postprandial state.
Changes in glucose status | Week 0 and 6
  Postprandial plasma samples are taken at the fasting state and 15, 30, 45, 60, 90, 120 and 180 min after consuming the study meal before, and after the 6-week diet intervention to see blood glucose development curve in postprandial state.
Changes in inflammation markers | Week 0 and 6
  The inflammation markers in plasma are measured as a baseline before the study and after 6 week diet intervention. The markers will be analysed with cDNA multiplex immunoassay and qPCR giving semi-quantitative results on a log2 scale (Olink inflammation panel, Olink Proteomics, Uppsala, Sweden). The panel contains at least 92 different proteins that are related to inflammation.
Changes in neuropsychological performance: cognitive load | Week 0 and 6
  Established and well-validated computerised neuropsychological tests to measure cognitive load will be conducted both at the beginning and at the end of the intervention in connection with postprandial test. Inquisit software (Millisecond Software, Seattle, Washington, USA; https://www.millisecond.com/download/library/) is used for the cognitive load (Serial Sevens Task) test.
Changes in neuropsychological performance: reaction time and attention | Week 0 and 6
  Established and well-validated computerised neuropsychological tests to measure cognitive load will be conducted both at the beginning and at the end of the intervention in connection with postprandial test. Inquisit software (Millisecond Software, Seattle, Washington, USA; https://www.millisecond.com/download/library/) is used for the reaction time and attention (Color Word Stroop test) test.
Changes in neuropsychological performance: response control | Week 0 and 6
  Established and well-validated computerised neuropsychological tests to measure cognitive load will be conducted both at the beginning and at the end of the intervention in connection with postprandial test. Inquisit software (Millisecond Software, Seattle, Washington, USA; https://www.millisecond.com/download/library/) is used for the response control (Cued Go/No-Go Task) test.

SECONDARY OUTCOMES:
Changes in gastrointestinal symptoms | Weeks 0 and 6
  Gastrointestinal symptoms (self-reported) during a postprandial study as measured by a questionnaire. The questionnaire is divided into seven types of gastrointestinal discomfort, and also includes a possibility to describe a gastrointestinal discomfort outside these seven given alternatives. The severity of the symptoms is self-reported on a three-step scale (0 as mild or no symptoms, 1 as moderate symptoms, 2 as strong symptoms).
Changes in gut microbiota | Week 0 and 6
  Changes in gut microbiota during the dietary intervention as seen in sequencing the fecal samples from the study participants before and after the 6-week dietary intervention.
Changes in excreted bile acids | Week 0 and 6
  Changes in excreted bile acids during the dietary intervention analyses from the fecal samples of the study participants before and after the 6-week dietary intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Food Sciences, Department of Life Technologies, University of Turku, Turku, Turku
  - Institute of Public Health and Clinical Nutrition, University of Eastern Finland, Kuopio

IPD SHARING:
Plan to Share IPD: Yes
Sensitive volunteer data may only be shared for collaborative research purposes with a separate agreement with the data owner. Metagenomic sequencing data can be found with identifier PRJEB104478 from ENA.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD will be available once the primary publications are published.
Access Criteria: Only for collaborative research purposes with a separate agreement with the data owner, the accessibility of data and documents can be decided together.